CLINICAL TRIAL: NCT02221713
Title: Assessment of the Gut Microbiome in Diverticulitis and Diverticulosis
Brief Title: The Gut Microbiome in Diverticulitis and Diverticulosis
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 163084
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Diverticulitis; Diverticulosis; Diverticular Disease
Keywords: diverticulitis; diverticulosis; diverticular disease
MeSH Terms: conditions — Diverticulitis; Diverticulum; Diverticular Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — stool samples and rectal swabs of stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group A: perforated diverticulitis: Patients with acute diverticulitis will be recruited from the A&E department at King's, prior to commencement of antibiotics. Rectal swabs will be obtained from patients with a chief complaint of acute abdominal pain upon initial assessment, prior to initial antibiotics. All specimens will be initially frozen, but only patients specimens with an admitting diagnosis of acute diverticulitis and colonic imaging (CT imaging or visualization at surgery) will be analysed. This group will include patients with perforated diverticulitis (i.e., Hinchey III or IV).
- Group B: unperforated diverticulitis: Patients with acute diverticulitis will be recruited from the A&E department at King's, prior to commencement of antibiotics. Rectal swabs will be obtained from patients with a chief complaint of acute abdominal pain upon initial assessment, prior to initial antibiotics. All specimens will be initially frozen, but only patients specimens with an admitting diagnosis of acute diverticulitis and colonic imaging (CT imaging or visualization at surgery) will be analysed. This group will include patients with unperforated diverticulitis (Hinchey I or II).
- Group C: asymptomatic diverticulosis: Patients with asymptomatic diverticulosis will be recruited from the 2-week wait (2ww) colorectal cancer pathway. Patients presenting with a chief complaint of fresh PR bleeding, with no other complaints, will be recruited prior to diagnostic imaging, either by CT, CT colonography, or endoscopy. They will provide a stool sample or rectal swab prior to bowel cleansing, if required for their evaluation, as that may alter the microbiome. Those patient samples with diverticulosis (and or haemorrhoids, as the other most common cause of fresh PR bleeding) will be analysed.
- Group D: normal controls: Patients with or without haemorrhoids, and no other colonic pathology will be recruited from the 2ww colorectal cancer pathway. These will be the normal controls. Patients presenting with a chief complaint of fresh PR bleeding, with no other complaints, will be recruited prior to diagnostic imaging, either by CT, CT colonography, or endoscopy. They will provide a stool sample or rectal swab prior to bowel cleansing, if required for their evaluation, as that may alter the microbiome. Those patient samples with diverticulosis (and or haemorrhoids, as the other most common cause of fresh PR bleeding) will be analysed.

SUMMARY:
Colonic diverticula are outpouchings of the large bowel, and they occur in up to 60% of people over 60 years of age. About 10-25% of patients with diverticula will have symptoms. These can range from acute diverticulitis, which can be a lethal infection to symptomatic diverticular disease, which involves inflammation of the bowel and altered bowel habits, decreasing patients' quality of life. We do not know which patients will develop acute diverticulitis or which patients will develop diverticula in their colon.

We believe that diverticulitis may be associated with, or even caused by, alterations in the bacteria that live in the colon, known as the gut microbiome. Until recently it was too expensive and too complex to examine the microbiome in detail. We propose to examine for the first time in detail the microbiome of patients with acute diverticulitis and asymptomatic diverticulosis.

Stool samples will be analysed for gut microbiome composition by 16S ribosomal RNA gene pyrosequencing. There is a part of the bacterial cell, the ribosome, which is the same in all bacteria (16S). Through PCR, polymerase chain reaction, and sequencing, we can separate out the different types of bacteria in a sample. We can then look at the different kinds of bacteria in each patient population, as well as how diverse the populations are within the groups, and compared to other groups.

We hope to be able to discriminate between the microbiome of patients with acute diverticulitis and asymptomatic diverticulosis. This study many change how diverticulitis and diverticulosis are conceptualized and treated. Alterations in the microbiome in these disease states may be able to be treated, preventing further disease.

DETAILED DESCRIPTION:
Diverticulosis affects 60% of people over 60 and roughly 10-25% of individuals will have symptoms, ranging from acute diverticulitis requiring emergent intervention to symptomatic diverticular disease with persistent lower abdominal pain and altered bowel habits. Up to 5% of patients with acute diverticulitis will die while hospitalized. In spite of the prevalence and severity of its manifestations, fundamental questions remain about the nature of diverticulitis and diverticulosis.

The human colon contains 100 trillion bacteria, including hundreds of species and 10 times as many genes as the human genome. While alterations in the microbiome have been implicated in disease states such as Irritable Bowel Syndrome (IBS) or Inflammatory Bowel Disease (IBD), the microbiome has not been adequately described in relation to colonic diverticula. As King's College Hospital has the only known dedicated Diverticular Disease clinic, we have a uniquely large patient population in which to learn about this condition.

When colonic diverticula become inflamed or perforate, patients have diverticulitis. Inciting factors for episodes of acute diverticulitis are not well characterized, but include age, lifestyle factors and certain medications. Clinicians have no way to predict which patients will get diverticulitis, nor how severe its presentation will be. In some cases of pericolonic diverticulitis (known as Hinchey I), inflammation may resolve even without antibiotics, while in other cases, perforated diverticulitis will include feculent peritonitis (Hinchey IV) and require emergent colon resection. Diverticulitis may be caused by alterations in the microbiome, but this has not been sufficiently addressed.

The majority of patients with asymptomatic diverticulosis, that is, the presence of colonic diverticula in the absence of symptoms, will never experience an episode of diverticulitis. There has been, however, some limited evidence that the microbiome in diverticulosis is altered, and similar to that in acute diverticulitis. If that is so, then predicting which patients will develop acute diverticulitis will remain impossible. It will also mean that research which did not assess or control for the presence of diverticula in patient populations will need to be revisited.

Currently, clinicians have no basis to predict (1) which patients will develop severe acute diverticulitis requiring surgery or (2) which patients will develop acute diverticulitis which will resolve with antibiotics. We believe that further insights into the gut microbiome will allow for better diagnostics and treatments in the future.

There have been a few, limited studies of the microbiome in diverticulitis, but not full pyrosequencing. This is because research costs have fallen 5 orders of magnitude in the past decade while computational capacity has increased. Studies have looked at the individual strains of bacteria within stool or mucosal samples, which does not suffice to understand the complex microbiome.

As the gut microbiome has not been thoroughly investigated in diverticular disease, this is an exploratory study. However, we do wish to test the hypotheses that patients with asymptomatic diverticulosis have a microbiome more similar to patients with acute diverticulitis, than to that of normal controls.

14. Methodology Setting: King's College Hospital, a tertiary referral hospital in south London. King's is a referral centre for the work up of two-week wait for colorectal cancer (2ww) assessments, with 900 new patient referrals assessed per year. Also, the Accident & Emergency Department at King's admits up to 250 patients per year with acute diverticulitis.

Patients: 4 sets of patients will be recruited. 25 patients per group will be recruited:

Groups A and B. Patients with acute diverticulitis will be recruited from the A&E department at King's, prior to commencement of antibiotics. Rectal swabs will be obtained from patients with a chief complaint of acute abdominal pain upon initial assessment, prior to initial antibiotics. All specimens will be initially frozen, but only patients specimens with an admitting diagnosis of acute diverticulitis and colonic imaging (CT imaging or visualization at surgery) will be analysed. Patients with acute diverticulitis will be assessed in 2 groups, those patients with perforated diverticulitis (i.e., Hinchey III or IV) and those patients with unperforated diverticulitis (Hinchey I or II).

Group C. Patients with asymptomatic diverticulosis will be recruited from the 2-week wait (2ww) colorectal cancer pathway. Patients presenting with a chief complaint of fresh rectal bleeding, with no other complaints, will be recruited prior to diagnostic imaging, either by CT, CT colonography, or endoscopy. They will provide a stool sample or rectal swab prior to bowel cleansing, if required for their evaluation, as that may alter the microbiome. Those patient samples with diverticulosis (and or haemorrhoids, as the other most common cause of fresh PR bleeding) will be analysed.

Group D. Patients with or without haemorrhoids, and no other colonic pathology will be recruited from the 2ww colorectal cancer pathway. These will be the normal controls. Patients presenting with a chief complaint of fresh PR bleeding, with no other complaints, will be recruited prior to diagnostic imaging, either by CT, CT colonography, or endoscopy. They will provide a stool sample or rectal swab prior to bowel cleansing, if required for their evaluation, as that may alter the microbiome. Those patient samples with diverticulosis (and or haemorrhoids, as the other most common cause of fresh PR bleeding) will be analysed.

Stool analysis: Stool samples will be analysed for faecal microbiome composition by 16S ribosomal RNA gene pyrosequencing, through a cooperative agreement with the Bruce lab at King's College London.

In brief, gene targeted 16S rRNA sequencing examines a structural component of the bacterial ribosome through targeted primers. Constant portions of the ribosomal RNA are amplified, which allows for identification of the variable portions. Sequences are then clustered in to OTUs, operational taxonomic units and may be assigned to lineages from genus all the way to phyla.

Planned statistical analyses: Microbiome composition will be assessed in several different ways. Alpha diversity will be measured, which is a measure of the average diversity within a sample. Multiple assessments of alpha diversity will be made, including Chaol richness estimate, OTU richness, and Shannon index. Alpha diversity has been shown to be reduced in patients with active IBD as compared to patients with quiescent disease, but has not been described in diverticular disease. Beta diversity is a comparison of diversity between samples (that is, the separation of the phylogenetic structure of the OTUs in one sample as compared to all other samples) will be calculated through Unifrac distances.

Power calculation: Metabonomic studies of the gut microbiome at this time are necessarily exploratory. As such power calculations have not been performed in the field. However, in this instance analysing 25 samples per group should be sufficient to discriminate between groups and assess their diversity.

Existing infrastructure: All infrastructure needed is currently in place. The study team (Professor Bjarnason and Mr Papagrigoriadis) currently manage the 2ww clinics, as well as attend to acute admissions in A&E at King's College Hospital. A materials transfer agreement is in place with the Bruce lab at King's College London for transfer of other faecal samples, and would only need to be amended.

ELIGIBILITY:
Inclusion Criteria:

Groups A and B. Patients with acute diverticulitis - patients presenting to A&E at King's College Hospital with new onset abdominal pain, with or without a known diagnosis of diverticulitis

Groups C and D. Patients with asymptomatic diverticulosis and normal controls

- Patients being assessed through the 2ww Colorectal Cancer pathway with a chief complaint of fresh PR bleeding and no other 'red flag' symptoms, who are not overly anxious over their diagnosis as assessed by a physician outside the study team.

Exclusion Criteria:

Groups A and B. Patients with acute diverticulitis

* Patients in extremis- e.g. systolic blood pressure less than 80 on arrival or pulse greater than 115
* Patients who have received antibiotics in the three months prior to presentation.
* Vulnerable patient populations

Groups C and D. Patients with asymptomatic diverticulosis and normal controls

* Patients with high levels of pre-test anxiety, as determined by their assessing physician, outside the study team
* Patients who received antibiotics for any reason in the 3 months prior to inclusion
* Vulnerable patient populations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Groups A and B. Patients with acute diverticulitis will be recruited from A&E at King's College Hospital. If they agree to participate, we will request either a stool sample to be produced, or, if that is not feasible, then a member of the study team will procure a rectal swab.
  Those patients with Hinchey III or IV's specimens will be assessed in Group A, while those patients with Hinchey I or II will be assessed in Group B.
  Groups C and D. Patients referred through the Two Week Wait (2ww) Colorectal Cancer pathway who are both at low risk for colorectal cancer and have low levels of anxiety, both as assessed by a physician outside the study team will be approached to participate. These patients will be able to produce the stool sample prior to presenting for flexible sigmoidoscopy as a part of their workup.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
assessment of gut microbiome | at time of enrollment
  Patients will give stool specimen or rectal swab after enrolling in the study. Stool samples will undergo 16S rRNA pyrosequencing for microbiome analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ingvar Bjarnason, MD, MSc FRCPath, FRCP(Glasg), Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, London, United Kingdom